CLINICAL TRIAL: NCT05878405
Title: Methylene Blue Mouthwash for Oral Mucositis Pain in Cancer: An Open-Label, Non-Randomized, Controlled Study
Brief Title: Methylene Blue Mouthwash for the Treatment of Oral Mucositis Pain in Patients With Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-007588; NCI-2023-03542 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-007588 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2023-05-10; First posted 2023-05-26 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm; Stomatitis
MeSH Terms: conditions — Stomatitis | interventions — Anti-Inflammatory Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Mouthwash Group (Active Comparator): Patients receive standard of care mouthwash as needed on study.
  Interventions: Other: Anti-inflammatory/Antimicrobial/Analgesic Aqueous Mouth Rinse
- Methylene Blue Mouthwash Group (Experimental): Patients receive Methylene Blue mouthwash as needed on study.
  Interventions: Other: Methylene Blue Oral Rinse

INTERVENTIONS:
Other: Anti-inflammatory/Antimicrobial/Analgesic Aqueous Mouth Rinse — Given PO
  Other Names: Dentoxol; Dentoxol Mouthrinse
  Arms: Standard of Care Mouthwash Group
Other: Methylene Blue Oral Rinse — Given PO
  Other Names: MB Oral Rinse
  Arms: Methylene Blue Mouthwash Group

SUMMARY:
This phase III trial compares the effect of methylene blue mouthwash to standard of care mouthwash for the treatment of oral mucositis pain in patients with cancer. Using methlylene blue mouthwash may improve oral pain in patients with oral mucositis related to cancer and/or cancer treatments compared to usual standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Active cancer diagnosis
* Admitted to the inpatient setting
* Pain related to oral mucositis
* Experiencing oropharyngeal pain
* Able to provide informed consent

Exclusion Criteria:

* Pediatric age (under 18 years old)
* Pregnant or nursing women
* Any contraindication to methylene blue including severe hypersensitivity to methylene blue and patients with glucose-6-phosphate dehydrogenase deficiency (G6PD) due to the risk of hemolytic anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Change in oral pain | Baseline, 3 days
  Pain will be assessed using the standard institutional numeric rating scale where pain level is quantified on a scale of 0 (no pain) to 10 (worst possible pain) pre- and post-intervention (3 times daily for 3 days). Last collected scores will be compared to baseline.

SECONDARY OUTCOMES:
Change in the amount of oral intake | Baseline, 3 days
  Electronic medical records will be reviewed for demographic and clinical information, medication administration record, and intake and output
Change in the amount of daily requirements of oral morphine equivalents | Baseline, 3 days
  Electronic medical records will be reviewed for demographic and clinical information, medication administration record, and intake and output

CONTACTS AND LOCATIONS:
Overall Officials: Regina M Mackey, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials